CLINICAL TRIAL: NCT04838340
Title: Effect of Hypnobirthing Training on Fear, Pain, Satisfaction Related to Birth and, Birth Outcomes: A Randomized Controlled Trial
Brief Title: Effect of Hypnobirthing Training on Fear, Pain, Satisfaction and, Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gonca Buran, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/GB
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Prenatal Education; Pregnancy Related; Labor Pain
Keywords: Childbirth; Labor Pain; Fear of childbirth; Satisfaction; Prenatal education; Hypnobirthing
MeSH Terms: conditions — Labor Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart care (Active Comparator): Standart care group will leave in the hospital's usual care and no intervention will be applied.
  Interventions: Other: Standart care
- Hypnobirthing group (Experimental): Hypnobirthig training intervention will be applied to the Hypnobirthing group for 4 weeks and 3 hours a week and usual care will be provided by healthcare professionals.
  Interventions: Behavioral: Hypnobirthig training

INTERVENTIONS:
Other: Standart care — This group will leave in the hospital's usual care and no intervention will be applied.
  Arms: Standart care
Behavioral: Hypnobirthig training — Hypnobirthing training of the Hypnobirthing group will carry out with its partner. Hypnobirthig training will be given in small groups of 5 or 6 couples for 4 weeks and 3 hours a week. In addition, the usual care will be provided by healthcare professionals to this group.
  Breathing, relaxation exercises, birth stories and birth videos will be used to reduce fears of chlildbirt women.
  Deepening and endorphin massage techniques will be given for labor pain. After the endorphin massage technique will be applied individually by the researcher, it will be applied by the couples and they will ask for repeating all exercises at home.
  In the last week of the training, there will be a birth rehearsal with Hynobirthing methods with the partners.
  The second meeting will take place when labor begins and after labor.
  Arms: Hypnobirthing group

SUMMARY:
Background and Purpose: Hypnobirthing is childbirth education model. This model aims for women to have a painless, calm and more comfortable birth. In this study is aimed to determine the effect of Hypnobirthing training on fear of childbirth, birth pain, birth satisfaction and birth outcomes.

Materials and Methods: This randomized controlled experimental study was performed in Maternity Hospital (Bursa, Turkey) . The minimum required sample size to be included in the study will calculated with G* power. The simple randomization method was use in the assignment of healthy and nulliparous pregnant women at 28-32 weeks of gestation to the groups. The assignment of the participants to the experimental group or control group was carried out with a computer-aided program. The nulliparous women was divided into two groups as the control group contained women who received the hospital's usual care, and the experimental group contained women who received the hypnobirthing training intervention. The fear of birth was measured with the Wijma Birth Expectancy/Experience Scale A and B (W-DEQ); labor pain was measured with Visual Analogue Scale (VAS); birth satisfaction was measured with Short Form of Birth Satisfaction Scale (BSS-R); birth outcomes will measure with postpartum Information form. The Statistical Package for the Social Sciences program (version 25.00) was use in data analysis.

DETAILED DESCRIPTION:
Fear of childbirth and labor pain are big problem that needs to be resolved as a priority since this situation continues by starting the vicious cycle of fear-anxiety-pain during childbirth. The persistence of the cycle increases the fear and pain related to childbirth, and thus delivery may result in emergency cesarean or elective cesarean. According to the data of Economic Development and Cooperation (OECD), the cesarean section rate in Turkey is 53.1% and so higher than the recommended rate, even Turkey has the highest rate among the OECD countries . High cesarean rates are an important problem that negatively affects maternal and infant health and increase health expenditures and costs. Therefore, the pregnant women education programs aimed at lowering the rate of cesarean section are still important in Turkey as in other countries. While the childbirth education programs for pregnant women are not widely practiced in Turkey, the Turkish Ministry of Health (TMOH) started to provide childbirth preparation courses to reduce the rate of cesarean section in recent years. In the circular issued by the TMOH in 2018, it was determined that these programs should be managed by physicians, obstetrics nurses, and midwives. Nurses are actively involved in pregnancy training programs where different methods are applied in Turkey as well as all over the world. The most common training methods applied in other countries are Lamaze Method, Bradly Method, and Hypnobirthing.

Hypnobirthing is a childbirth preparation method that aims to prepare pregnant women for delivery mentally and physically and to give birth in a less painful, conscious, and fear-free way. This method was developed based on the fear-stress-pain cycle. The persistence of this cycle exacerbates stress and pain, prolongs the birth period, and negatively affects the success, way, preference, course, and satisfaction of the birth. Thus, the birth does not proceed properly and results in an emergency or elective cesarean section. Hypnobirthing can prepare women for childbirth to eliminate all these negativities.

Hypnobirthing training can be considered as a new technique for Turkey and therefore we conducted this study to determine its effects on the pain, fear, satisfaction related to childbirth and childbirth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primiparas
* Ages between 18-42
* In gestational week 28-32
* Being literate in Turkish
* Pregnant with a single child
* Minimum a primary school graduate (since the questionnaires would be filled out by self-reporting)

Exclusion Criteria:

* High-risk pregnancy (on the basis of the criteria of the Ministry of Health)
* Attended other prenatal training sessions (pregnancy pilates and yoga)
* High-risk pregnancy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 80 (Actual)
Dates: Start 2019-05-04 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
Preinterventional Scores on the W-DEQ-A (the minimum values:0, maximum:165) | When the control and experimental groups were Enrollment in the study
  Distribution of the scores of pregnant women on the W-DEQ-A before the intervention to the experimental and control groups. Higher scores are worse outcome.
The VAS scores of the experimental and control groups (the minimum values:0, maximum=10) | in the process of labor (the first stage of labor: latent, active and transitional phases )
  Distribution of the women on the VAS in the first stage of labor according to the experimental and control groups. Higher scores are worse outcome.
W-DEQ-B Scores (the minimum values:0, maximum:160) | within eight hours after birth
  Distribution of the scores of the women on the whole W-DEQ-B according to the control and experimental groups. Higher scores are worse outcome.
The chilbirth scores of the experimental and control groups (questionnaire) | within eight hours after birth
  Information about the childbirth of the experimental and control groups ( childbirth position, Intervention at birth, way of delivery, duration of delivery)
BSS-R scores of experimental and control groups (the minimum values:0, maximum:40) • Low level of satisfaction ˂13 points, • Medium satisfaction level 14-27 points, • High satisfaction level ≥28 | within eight hours after birth
  Postpartum scores of the control and experimental groups on the BSS-R. Higher scores are better outcome.

SECONDARY OUTCOMES:
Women and baby interaction | within eight hours after birth
  The first skin to skin contact time and the first breastfeeding time of the women in the control and experimental groups

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Buran, PhD, Principal Investigator — Uludag Üniversity; Hilmiye Aksu, Professor, Study Director — Adnan Menderes Üniversity
Locations (1):
- Gonca Buran, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no a plan to make individual participant data (IPD) available to other researcher on Clinical Trails.cov.

REFERENCES:
- [Background] Varner CA. Comparison of the Bradley Method and HypnoBirthing Childbirth Education Classes. J Perinat Educ. 2015;24(2):128-36. doi: 10.1891/1946-6560.24.2.128. PMID 26957896
- [Background] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- [Background] Saisto T, Halmesmaki E. Fear of childbirth: a neglected dilemma. Acta Obstet Gynecol Scand. 2003 Mar;82(3):201-8. PMID 12694113
- [Background] Korukcu O, Kukulu K, Firat MZ. The reliability and validity of the Turkish version of the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) with pregnant women. J Psychiatr Ment Health Nurs. 2012 Apr;19(3):193-202. doi: 10.1111/j.1365-2850.2011.01694.x. Epub 2012 Jan 20. PMID 22260727
- [Background] Hollins Martin CJ, Martin CR. Development and psychometric properties of the Birth Satisfaction Scale-Revised (BSS-R). Midwifery. 2014 Jun;30(6):610-9. doi: 10.1016/j.midw.2013.10.006. Epub 2013 Oct 24. PMID 24252712
- [Background] Goncu Serhatlioglu S, Karahan N, Hollins Martin CJ, Martin CR. Construct and content validity of the Turkish Birth Satisfaction Scale - Revised (T-BSS-R). J Reprod Infant Psychol. 2018 Jul;36(3):235-245. doi: 10.1080/02646838.2018.1443322. Epub 2018 Mar 19. PMID 29553295
- [Background] Sercekus P, Okumus H. Fears associated with childbirth among nulliparous women in Turkey. Midwifery. 2009 Apr;25(2):155-62. doi: 10.1016/j.midw.2007.02.005. Epub 2007 Jun 27. PMID 17600599
- [Result] Fenwick J, Toohill J, Gamble J, Creedy DK, Buist A, Turkstra E, Sneddon A, Scuffham PA, Ryding EL. Effects of a midwife psycho-education intervention to reduce childbirth fear on women's birth outcomes and postpartum psychological wellbeing. BMC Pregnancy Childbirth. 2015 Oct 30;15:284. doi: 10.1186/s12884-015-0721-y. PMID 26518597
- [Result] Phillips-Moore J. HypnoBirthing. Aust J Holist Nurs. 2005 Apr;12(1):41-2. No abstract available. PMID 19175270
- [Result] Kobayashi S, Hanada N, Matsuzaki M, Takehara K, Ota E, Sasaki H, Nagata C, Mori R. Assessment and support during early labour for improving birth outcomes. Cochrane Database Syst Rev. 2017 Apr 20;4(4):CD011516. doi: 10.1002/14651858.CD011516.pub2. PMID 28426160
- [Result] Hodnett ED, Gates S, Hofmeyr GJ, Sakala C. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2013 Jul 15;7:CD003766. doi: 10.1002/14651858.CD003766.pub5. PMID 23857334